CLINICAL TRIAL: NCT04199169
Title: A Phase 1 Randomized, Placebo-controlled, Observer-blind Trial to Assess the Safety and Immunogenicity of a Nipah Vaccine, HeV-sG-V (Hendra Virus Soluble Glycoprotein Vaccine), in Healthy Adults
Brief Title: Safety and Immunogenicity of a Nipah Virus Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Auro Vaccines LLC (Industry)
Collaborators: PATH (Other); Coalition for Epidemic Preparedness Innovations (Other); Cincinnati Children's Hospital Medical Center (CCHMC) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CVIA 077; HeV-sG-01
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Nipah Virus Infection
Keywords: Nipah, Vaccine, Henipah
MeSH Terms: conditions — Henipavirus Infections

STUDY DESIGN:
Intervention Model Description: Ascending dose study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1, Group 1 (Experimental): Ten subjects in the first cohort will receive a 10 mcg dose of HeV-sG-V on Visits 1 and 6.5 (Days 1 and 169*).
  *Second dose was administered at 6 months due to study pause from local COVID-19 shutdown.
  Interventions: Biological: HeV-sG-V
- Cohort 1, Group 2 (Placebo Comparator): Two subjects in the first cohort will receive a dose of the placebo on Visits 1 and 6.5 (Days 1 and 169*).
  *Second dose was administered at 6 months due to study pause from local COVID-19 shutdown.
  Interventions: Biological: Normal Saline Placebo
- Cohort 2, Group 3 (Experimental): Thirty subjects in the second cohort will receive a 30 mcg dosage of HeV-sG-V on Visits 1 and 2 (Days 1 and 8) with placebo on Visit 3 (Day 29).
  Interventions: Biological: HeV-sG-V; Biological: Normal Saline Placebo
- Cohort 2, Group 4 (Experimental): Thirty subjects in the second cohort will receive a 30 mcg dosage of HeV-sG-V on Visits 1 and 3 (Days 1 and 29) with placebo on Visit 2 (Day 8)
  Interventions: Biological: HeV-sG-V; Biological: Normal Saline Placebo
- Cohort 2, Group 5 (Placebo Comparator): Twelve subjects in the second cohort will receive a dose of the placebo on Visits 1, 2, and 3 (Days 1, 8 and 29).
  Interventions: Biological: Normal Saline Placebo
- Cohort 3, Group 6 (Experimental): Thirty subjects in the third cohort will receive a 100 mcg dosage of HeV-sG-V on Visit 1 (Day 1) and placebo on Visits 2 and 3 (Days 8 and 29).
  Interventions: Biological: HeV-sG-V; Biological: Normal Saline Placebo
- Cohort 3, Group 7 (Experimental): Thirty subjects in the third cohort will receive a 100 mcg dosage of HeV-sG-V on Visits 1 and 2 (Days 1 and 8) and placebo on Visit 3 (Day 29).
  Interventions: Biological: HeV-sG-V; Biological: Normal Saline Placebo
- Cohort 3, Group 8 (Experimental): Thirty subjects in the third cohort will receive a 100 mcg dosage of HeV-sG-V on Visits 1 and 3 (Days 1 and 29) and placebo on Visit 2 (Day 8).
  Interventions: Biological: HeV-sG-V; Biological: Normal Saline Placebo
- Cohort 3, Group 9 (Placebo Comparator): Eighteen subjects in the third cohort will receive a dose of the placebo on Visits 1, 2, and 3 (Days 1, 8 and 29).
  Interventions: Biological: Normal Saline Placebo

INTERVENTIONS:
Biological: HeV-sG-V — A Hendra virus soluble glycoprotein vaccine formulated in phosphate buffer and adjuvanted with aluminum hydroxide. Placebo is normal saline.
  Other Names: Nipah Vaccine, HenipaVaxTM
  Arms: Cohort 1, Group 1; Cohort 2, Group 3; Cohort 2, Group 4; Cohort 3, Group 6; Cohort 3, Group 7; Cohort 3, Group 8
Biological: Normal Saline Placebo — 0.9% Saline
  Other Names: Placebo
  Arms: Cohort 1, Group 2; Cohort 2, Group 3; Cohort 2, Group 4; Cohort 2, Group 5; Cohort 3, Group 6; Cohort 3, Group 7; Cohort 3, Group 8; Cohort 3, Group 9

SUMMARY:
A first-in-human, phase 1 trial is to be conducted in a healthy adult population in the US to assess the safety and immunogenicity of three ascending Nipah vaccine (HeV-sG-V; Hendra virus soluble glycoprotein vaccine) dosages. Different dosing regimens and number of doses will also be explored.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, observer-blind, phase 1 trial in healthy male and non-pregnant female adults 18 through 49 years of age designed to assess the safety and immunogenicity of three ascending doses of HeV-sG-V. Different dosing regimens and number of doses will also be explored.

The study plans to accrue eligible subjects into three successive dosage escalation cohorts consisting of 12, 72, and 108 subjects, respectively (total of 192 subjects). The three HeV-sG-V dosages will be 10 mcg, 30 mcg, and 100 mcg.

In the first cohort, subjects will receive two doses of the investigational product (IP) at 28-day intervals. Subjects will be randomized in a 5:1 ratio, with 10 receiving two doses of HeV-sG-V (10 mcg dosage) and two subjects will receive placebo.

In the second cohort, subjects will be randomized in a 5:5:2 ratio with 30 receiving a 30 mcg dosage of HeV-sG-V on Visits 1 and 2 (Days 1 and 8) with placebo on Visit 3 (Day 29), 30 receiving a 30 mcg dosage of HeV-sG-V on Visits 1 and 3 (Days 1 and 29) with placebo on Visit 2 (Day 8), while 12 subjects will receive placebo at each of the same visits.

The third cohort will be randomized in a 5:5:5:3 ratio so that 30 subjects are assigned to each of three different regimens consisting of a 100 mcg dosage of HeV-sG-V and placebo administered as three doses, HeV-sG-V on Visit 1 (Day 1) with placebo on Visits 2 and 3 (Days 8 and 29), or HeV-sG-V on Visits 1 and 2 (Days 1 and 8) with placebo on Visit 3 (Day 29), or HeV-sG-V on Visits 1 and 3 (Days 1 and 29) with placebo on Visit 2 (Day 8), while the remaining 18 will receive a dose of placebo at each of the same visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female 18 through 49 years of age at the time of consenting and IP administration.
2. Provides written informed consent prior to performance of any study-specific procedure.
3. Resides in study site area and is able and willing to adhere to all protocol visits and procedures, including plasmapheresis.
4. Healthy, as defined by absence of any clinically significant medical conditions, either acute or chronic, as determined by medical history, physical examination, safety laboratory test results, and clinical assessment of the investigator.
5. Female subjects of childbearing potential* must have practiced adequate contraception** for 28 days prior to administration of IP and agree to continue adequate contraception until completion of the plasmapheresis session or Visit 5 (Day 57) for subjects not selected for plasmapheresis.

   * Females can be considered not of childbearing potential if they are with current bilateral tubal ligation or occlusion, or post-hysterectomy, or post-bilateral ovariectomy, or post-menopause.

   ** Adequate contraception is defined as a contraceptive method with failure rate of less than 1% per year when used consistently and correctly and when applicable, in accordance with the product label, for example:
   * Abstinence from penile-vaginal intercourse
   * Combined estrogen and progesterone oral contraceptives
   * Injectable progestogen
   * Implants of etonogestrel or levonorgestrel
   * Contraceptive vaginal ring
   * Percutaneous contraceptive patches
   * Intrauterine device or intrauterine system
   * Male condom combined with a vaginal spermicide (foam, gel, film, cream or suppository), and/or progesterone alone oral contraceptive
6. Female subjects of childbearing potential must have a negative pregnancy test within 24 hours prior to IP administration.

Exclusion Criteria:

1. Previous immunization with an investigational Nipah or Hendra virus vaccine.
2. History of disease known to be caused by Nipah or Hendra virus.
3. Travel to Kerala state, India within the previous three years or planned travel to Kerala sate or Bangladesh during the study period.
4. Known hypersensitivity to any component of the IPs.
5. Known hypersensitivity to citrate or ethylene oxide.
6. History of hypersensitivity to any vaccine.
7. Administration of any vaccine other than the IP within 28 days prior to IP administration or planned administration through completion of plasmapheresis or Visit 5 (Day 57) for subjects not selected for plasmapheresis.
8. Administration of any investigational or non-registered drug within 90 days prior to IP administration or planned administration during the study period.
9. Administration of immunoglobulin or any blood product within 90 days prior to IP administration or planned administration during the study period.
10. Administration of any long-acting immune-modifying drugs (e.g., infliximab or rituximab) or the chronic administration (defined as more than 14 days) of immunosuppressants within 180 days prior to IP administration or planned administration during the study period (includes systemic corticosteroids at doses equivalent to ≥ 0.5 mg/kg/day of prednisone; topical steroids including inhaled and intranasal steroids are not exclusionary).
11. Acute illness or fever (body temperature measured orally ≥ 38°C or 100.4°F) at the time of IP administration (once acute illness/fever is resolved, if appropriate, as per investigator assessment, subject may be screened again).
12. History of or evidence for chronic clinically significant (as per investigator assessment) disorder or disease (including, but not limited to immunodeficiency, autoimmunity, bleeding or psychiatric disorder, and pulmonary, cardiovascular, metabolic, neurologic, renal, or hepatic disease).
13. Any condition that in the opinion of the investigator might compromise the safety or well-being of the subject or compromise adherence to protocol procedures or interfere with planned safety and immunogenicity assessments.
14. History of chronic alcohol consumption or drug abuse that in the opinion of the investigator might compromise adherence to protocol procedures or interfere with planned safety and immunogenicity assessments.
15. Blood donation or planned blood donation within 28 days prior to IP administration through 28 days after completion of the plasmapheresis session or Visit 5 (Day 57) for subjects not selected for plasmapheresis.
16. Pregnant.
17. Body weight < 50 kg.
18. Body Mass Index (BMI) ≥ 40 kg/m2.
19. Infection with human immunodeficiency virus 1 or 2.
20. Infection with hepatitis B or hepatitis C virus.
21. The following clinical safety laboratory test results will be considered exclusionary, regardless of assessment of clinical significance:

Hemoglobin (Male) < 13.3 g/dL Hemoglobin (Female) < 12.8 g/dL Hematocrit > 55% Neutrophil count < 1,500 cells/mm3 Eosinophil count > 600 cells/mm3 Platelet count < 130,000 cells/mm3 Creatinine > 1.4 mg/dL ALT > 1.1 x upper limit of the normal range (ULN)* [* per the site clinical laboratory's reference ranges]

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Rate of local and systemic solicited adverse events | for 1 week after each innoculation
  e.g., headache, fatigue, fever, etc.that are specifically asked about by the doctor
Incidence of clinically significant abnormalities in clinical safety laboratory test results reported as unsolicited AEs. | for 1 week after each innoculation
  e.g. hemoglobin, white blood cell count, neutrophil count, creatinine, etc.
Incidence of unsolicited adverse events | for 1 month after the last vaccination
  Adverse events that are reported to the doctor beyond what is asked about by the doctor. An adverse event is any undesirable experience associated with the use of a medical product in a patient.
Incidence of medically attended adverse events and serious adverse events | through Day 197
  A reaction to the vaccine that require medical attention. Serious adverse events can include death, hospitalization, disability, and death.

SECONDARY OUTCOMES:
Determine number of doses and timing of doses required | through day 57
  Quantitative measurement of antibody response to virus
Determine number of doses and timing of doses required | through day 57
  Qualitative measurement of antibody response to virus

CONTACTS AND LOCATIONS:
Overall Officials: Robert W. Frenck Jr., MD, Principal Investigator — Cincinnati Children's Hospital Medical Center (CCHMC)
Locations (1):
- Cincinnati Children's Hospital Medical Center (CCHMC), Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No